CLINICAL TRIAL: NCT04136093
Title: Defining the Optimal Dietary Strategy for the Maintenance of Weight Loss and mEtaboLiC Outcomes in Centrally Obese postMenopausal womEn (WELCOME Study).
Brief Title: Diet for the Maintenance of Weight Loss and Metabolic Health in Obese Postmenopausal Women
Acronym: WELCOME
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Poznan University of Life Sciences (Other)
Responsible Party: Principal Investigator, Lidia Małczak, Principal Investigator, Poznan University of Life Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 445446
Record Dates: First submitted 2019-10-21; First posted 2019-10-23 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Metabolic Syndrome; Diet Modification; Postmenopause
Keywords: Weight Loss Maintenance; Metabolic Disorders; Postmenopausal Women; Cardiometabolic Parameters; Diet Therapy; Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome; Metabolic Diseases

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- the MED (Experimental): The 50 postmenopausal women who in phase I will lose ≥10% of initial body weight will be randomly assigned to the MED group
  Interventions: Other: the MED
- the DASH (Experimental): The 50 postmenopausal women who in phase I will lose ≥10% of initial body weight will be randomly assigned to the DASH group
  Interventions: Other: the DASH
- The control group (Experimental): The 50 postmenopausal women who in phase I will lose ≥10% of initial body weight will be randomly assigned to the control group.
  Interventions: Other: Control diet

INTERVENTIONS:
Other: the MED — The MED diet will be composed of the basis food items traditional for the Mediterranean region i.e. olive oil, nuts, vegetables, fruits, and fish and this diet will be given an ad libitum approach. The MED diet will be giving a higher proportion of fat, at least 40% of the total energy, with 20% of the total energy from MUFAs, and less proportion of carbohydrates. To ensure the assumed supply of MUFAs and polyunsaturated fatty acids (PUFAs), the participants will be asked to daily intake 60 g (6 spoons) of extra virgin olive oil and 30 g (6 pieces) walnuts.
  Arms: the MED
Other: the DASH — The DASH diet will be giving a higher proportion of carbohydrates, at least 60% of total energy and less fat. The DASH diet will be composed wholegrain cereal products, fruit, vegetables, low-fat dairy products, fish, seafood, poultry, beans, seeds and nuts and will be recommending eating of the traditional polish food items for example oatmeal, rye bread, barley groats, apples, plums, etc. and reducing the supply of salt, sweets, sugars, fats especially saturated fats and red meat. In our study, the DASH diet will be given an ad libitum approach. The sufficient supply of carbohydrates and β glucans in the DASH diet will be ensured by daily consumption at least 50g oatmeal and 50g of barley groats.
  Arms: the DASH
Other: Control diet — The control group will only receive oral dietary recommendations based on the Harvard model "Healthy Eating Plate", that recommend to eat a half of plate of vegetables and fruit, a quarter of plate of whole grains products, and a quarter of plate of protein products for one meal.
  Arms: The control group

SUMMARY:
The aim of the study will be comparing the effectiveness of two diets: moderate in fat with a high proportion of monounsaturated fatty acids (MUFAs) - the Mediterranean diet (MED) and 2) the low in fat and high in dietary fiber contents the dietary approaches to stop hypertension diet (DASH) on weight maintenance and cardiovascular risks following a recent body weight reduction in centrally obese postmenopausal women. The tested diets will be given ad libitum manner. Moreover, adherence to both prescribed weight-loss maintenance diets will be also evaluated by the plasma concentration of alkylresorcinols (AR) as a possible whole grain wheat/rye dietary biomarker and by the analysis of fatty acids profile in erythrocyte membranes as a dietary biomarker of a fatty acids consumption. The participants of this study will be 150 non-smoking, postmenopausal women with central obesity, who wished to lose weight and have at least one other criterion of metabolic syndrome. The intervention will include 3 phases: Phase I (weeks 1-8), weight loss dietary intervention with 700 kcal/d energy deficit, Phase II (week 9-32), weight loss maintenance intervention for those participants losing ≥10% initial body weight the MED or the DASH diet will be offered in a random manner. The control group will receive oral dietary recommendations based on the Harvard model "Healthy Eating Plate". After this 32 weeks period will be finished, the participants will be discharged to the community with no contact by study personnel, until the 52-weeks follow-up period (Phase III).

DETAILED DESCRIPTION:
The treatment of obesity can present a challenge because of the difficulty in maintaining body weight loss beyond one year. The aim of the study will be comparing the effectiveness of two energy-unrestricted diets containing different amount of macronutrients: 1) moderate in fat with high amounts of MUFAs - the MED diet and 2) low in fat with high dietary fiber contents - the DASH diet, on maintenance of weight loss and metabolic outcomes following a recent weight loss in centrally obese postmenopausal women. Since the outcomes of dietary interventions may depend greatly on adherence to the diet, we will measure the plasma AR concentrations and fatty acids profile in red blood cells (RBC). Plasma AR concentrations is a valid marker of intake of whole-grain wheat/rye in the DASH diet and fatty acids concentration in RBC is a valid marker of fatty acids intake (especially MUFAs) in the MED diet. A total of 150 non-smoking, centrally obese, with at least one other criterion of metabolic syndrome postmenopausal women up to 65 old years will be qualified. This study will be divided into 3 phases:

* Phase I lasting eight weeks (weeks 1-8). All participants will be introduced to a weight loss intervention with a daily energy deficit of 700 kcal per day. During this phase, changes in body weight and body composition (DEXA) and waist circumference will be measured every four weeks. Moreover, at each control visit, compliance with the prescribed diets will be measured by three-day food records. Moreover, the physical activity level will be done. Before and after weight loss phase changes in lipid and non-lipid parameters as well as eating behavior will be measured.
* Participants who will loss ≥10% initial body weight will be randomly assigned to phase II of the study (weight loss maintenance intervention). This phase will be lasting 24 weeks (weeks 9-32). Participants will receive the MED (n = 50) or DASH diet (n = 50). The control group (n = 50) will receive oral dietary recommendations based on the Harvard model "Healthy Eating Plate". During this phase, changes in body weight, body composition, and waist circumference will be measured every four weeks. Moreover, at each control visit, compliance with the prescribed diets will be measured by three-day food records. Moreover, the physical activity level will be done. Before and after weight loss phase changes in lipid and non-lipid parameters as well as valid markers of whole-grain wheat/rye and faty acids intake and eating behavior will be measured.
* After this 32 weeks period will be finished, the participants will be discharged to the community with no contact from study personnel for 20 weeks, until follow-up at 52 weeks study (Phase III - weeks 33 - 52). After this time changes in body weight, body composition and waist circumference will be measured. Moreover, the physical activity level will be done again and changes in lipid and non-lipid parameters, as well as valid markers of intake and eating behavior, will be measured.

ELIGIBILITY:
Inclusion Criteria:

* postmenopausal women, with the absence of menses of over 12 months or serum follicle stimulating hormone > 30 IU/mL;
* with central obesity waist circumference (WC) ≥ 80 cm
* with low physical activity (PAL = 1,40);
* who wished to lose weight and weight loss maintenance;
* and have at least one other criterion of metabolic syndrome increased systolic blood pressure ≥ 130 mm Hg or high blood pressure diastolic ≥ 85 mm Hg or ongoing treatment of previously diagnosed hypertension, increased serum triglyceride levels above >150 mg/dl (1.7 mmol/l) or ongoing therapy hypertriglyceridemia, decreased HDL cholesterol below than <50 mg/dl (1.3 mmol/l), and fasting blood glucose > 100 mg/dl (5.6 mmol / l) or ongoing treatment of previously diagnosed type 2 diabetes.

Exclusion Criteria:

* thyroid disease (hypothyroidism, hyperthyroidism, thyroiditis);
* hypercortisolism, Cushing's syndrome;
* kidney diseases;
* type 1 diabetes;
* asthma treated with oral and injectable steroids;
* cancers; mental disorders;
* New York Heart Association (NYHA) Class III heart failure;
* as well as any drug is known to influence liver function;
* endocrine disorders;
* hormonal replacement therapy;
* significant weight change in the six months prior to the current study;
* impaired absorption of nutrients (celiac disease, inflammatory bowel disease);
* intolerance or food allergy to key components of the intervention diets;
* smoking
* excessive alcohol consumption (consumption of more than 2 alcohol units per day - one alcohol unit equals one bottle of beer (340 g) or one glass of wine (140 g) or one glass of spirits (42.5 g of 40% spirit).

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Postmenopausal women, with the absence of menses of over 12 months or serum follicle stimulating hormone > 30 IU/mL.
Enrollment: 150 (Estimated)
Dates: Start 2020-02-29 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Changes in body weight [kg] | measurements will be taken after 8 weeks of weight loss diet (before weight loss maintenance period) and after 12, 16, 20, 24, 28, 32 and after 52 week of study.
  Changes in body weight from 9 to 52 week of weight loss maintenance period
Changes in waist circumferences (WC) [cm] | measurements will be taken after 8 weeks weight loss diet (before weight loss maintenance period) and after 12, 16, 20, 24, 28, 32 and after 52 week of study.
  Changes in waist circumferences from 9 to 52 week of weight loss maintenance period.
Changes in fat mass [kg] | measurements will be taken after 8 weeks weight loss diet (before weight loss maintenance period) and after 12, 16, 20, 24, 28, 32 and after 52 week of study.
  Changes in fat mass from 9 to 52 weeks of weight loss maintenance period.
Changes in HDL cholesterol [mg/dL] | Examination will be taken after 8 weeks weight loss diet (before weight loss maintenance period) after 32 and also after 52 week of study.
  Changes in HDL cholesterol from 9 to 52 week of weight loss maintenance period.
changes in triglycerides (TG) [mg/dL] | Examination will be taken after 8 weeks weight loss diet (before weight loss maintenance period) after 32 and also after 52 week of study.
  Changes in TG from 9 to 52 week of weight loss maintenance period.
changes in glucose (GLU) | Examination will be taken after 8 weeks weight loss diet (before weight loss maintenance period) after 32 and 52 week of study.
  Changes in GLU from 9 to 52 week of weight loss maintenance period.
Changes in systolic blood pressure (SBP) | measurements will be taken after 8 weeks weight loss diet (before weight loss maintenance period) and after 12, 16, 20, 24, 28, 32 and also after 52 week of study.
  Changes in SBP from 9 to 52 week of weight loss maintenance period.
Changes in diastolic blood pressure (DBP) | measurements will be taken after 8 weeks weight loss diet (before weight loss maintenance period) and after 12, 16, 20, 24, 28, 32 and also after 52 week of study.
  Changes in DBP from 9 to 52 weeks of weight loss maintenance period.

SECONDARY OUTCOMES:
Physical activity level (PAL) | The assessment of the PA level will be done after 8 weeks of weight loss diet (before weight loss maintenance period) and after 32 and 52 week of study.
  The assessment of the PAL from 9 to 52 week weight loss maintenance period.
Eating behaviour (by measurement of dietary restraint, disinhibition and hunger) | The assessment of the eating behaviour will be done after 8 weeks of weight loss diet (before weight loss maintenance period), after 32 and also after 52 week of study.
  The assessment of the eating behaviour from 9 to 52 week weight loss maintenance period.
Adherence to the prescribed diets (assessment of the plasma AR levels and concentration and fatty acids in red blood cells) | The assessment of the adherence will be done after 12, 16, 20, 24, 28 and 32 week of study.
  The assessment of the adherence from 9 to 32 weeks weight loss maintenance period.
Dietary intake | Each participant"s dietary records will be assessed after 12, 16, 20, 24, 28, and 32 and also after 52 week of study.
  The assessment of the dietary intake from 9 to 52 weeks weight loss maintenance period.

CONTACTS AND LOCATIONS:
Overall Officials: Lidia Małczak, MSc, Principal Investigator — Poznań University of Life Sciences
Locations (1):
- Poznan University of Life Science, Poznan, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bajerska J, Chmurzynska A, Muzsik A, Krzyzanowska P, Madry E, Malinowska AM, Walkowiak J. Weight loss and metabolic health effects from energy-restricted Mediterranean and Central-European diets in postmenopausal women: A randomized controlled trial. Sci Rep. 2018 Jul 24;8(1):11170. doi: 10.1038/s41598-018-29495-3. PMID 30042488
- [Background] Beavers DP, Beavers KM, Lyles MF, Nicklas BJ. Cardiometabolic risk after weight loss and subsequent weight regain in overweight and obese postmenopausal women. J Gerontol A Biol Sci Med Sci. 2013 Jun;68(6):691-8. doi: 10.1093/gerona/gls236. Epub 2012 Nov 26. PMID 23183902
- [Background] Beunza JJ, Toledo E, Hu FB, Bes-Rastrollo M, Serrano-Martinez M, Sanchez-Villegas A, Martinez JA, Martinez-Gonzalez MA. Adherence to the Mediterranean diet, long-term weight change, and incident overweight or obesity: the Seguimiento Universidad de Navarra (SUN) cohort. Am J Clin Nutr. 2010 Dec;92(6):1484-93. doi: 10.3945/ajcn.2010.29764. Epub 2010 Oct 20. PMID 20962161
- [Background] Elfhag K, Rossner S. Who succeeds in maintaining weight loss? A conceptual review of factors associated with weight loss maintenance and weight regain. Obes Rev. 2005 Feb;6(1):67-85. doi: 10.1111/j.1467-789X.2005.00170.x. PMID 15655039
- [Background] FOLCH J, LEES M, SLOANE STANLEY GH. A simple method for the isolation and purification of total lipides from animal tissues. J Biol Chem. 1957 May;226(1):497-509. No abstract available. PMID 13428781
- [Background] Gibson AA, Sainsbury A. Strategies to Improve Adherence to Dietary Weight Loss Interventions in Research and Real-World Settings. Behav Sci (Basel). 2017 Jul 11;7(3):44. doi: 10.3390/bs7030044. PMID 28696389
- [Background] Hedrick VE, Dietrich AM, Estabrooks PA, Savla J, Serrano E, Davy BM. Dietary biomarkers: advances, limitations and future directions. Nutr J. 2012 Dec 14;11:109. doi: 10.1186/1475-2891-11-109. PMID 23237668
- [Background] Hernaez A, Castaner O, Elosua R, Pinto X, Estruch R, Salas-Salvado J, Corella D, Aros F, Serra-Majem L, Fiol M, Ortega-Calvo M, Ros E, Martinez-Gonzalez MA, de la Torre R, Lopez-Sabater MC, Fito M. Mediterranean Diet Improves High-Density Lipoprotein Function in High-Cardiovascular-Risk Individuals: A Randomized Controlled Trial. Circulation. 2017 Feb 14;135(7):633-643. doi: 10.1161/CIRCULATIONAHA.116.023712. PMID 28193797
- [Background] Kozakowski J, Gietka-Czernel M, Leszczynska D, Majos A. Obesity in menopause - our negligence or an unfortunate inevitability? Prz Menopauzalny. 2017 Jun;16(2):61-65. doi: 10.5114/pm.2017.68594. Epub 2017 Jun 30. PMID 28721132
- [Background] Krishnan S, Cooper JA. Effect of dietary fatty acid composition on substrate utilization and body weight maintenance in humans. Eur J Nutr. 2014 Apr;53(3):691-710. doi: 10.1007/s00394-013-0638-z. Epub 2013 Dec 22. PMID 24363161
- [Background] Sacks FM, Bray GA, Carey VJ, Smith SR, Ryan DH, Anton SD, McManus K, Champagne CM, Bishop LM, Laranjo N, Leboff MS, Rood JC, de Jonge L, Greenway FL, Loria CM, Obarzanek E, Williamson DA. Comparison of weight-loss diets with different compositions of fat, protein, and carbohydrates. N Engl J Med. 2009 Feb 26;360(9):859-73. doi: 10.1056/NEJMoa0804748. PMID 19246357
- [Background] Santoro N. The menopausal transition. Am J Med. 2005 Dec 19;118 Suppl 12B:8-13. doi: 10.1016/j.amjmed.2005.09.008. PMID 16414322
- [Background] Soeliman FA, Azadbakht L. Weight loss maintenance: A review on dietary related strategies. J Res Med Sci. 2014 Mar;19(3):268-75. PMID 24949037
- [Background] Stachowiak G, Pertynski T, Pertynska-Marczewska M. Metabolic disorders in menopause. Prz Menopauzalny. 2015 Mar;14(1):59-64. doi: 10.5114/pm.2015.50000. Epub 2015 Mar 25. PMID 26327890
- [Background] Thom G, Lean M. Is There an Optimal Diet for Weight Management and Metabolic Health? Gastroenterology. 2017 May;152(7):1739-1751. doi: 10.1053/j.gastro.2017.01.056. Epub 2017 Feb 15. PMID 28214525
- [Background] Desroches S, Lapointe A, Ratte S, Gravel K, Legare F, Turcotte S. Interventions to enhance adherence to dietary advice for preventing and managing chronic diseases in adults. Cochrane Database Syst Rev. 2013 Feb 28;2013(2):CD008722. doi: 10.1002/14651858.CD008722.pub2. PMID 23450587
- [Background] Yannakoulia M, Kontogianni M, Scarmeas N. Cognitive health and Mediterranean diet: just diet or lifestyle pattern? Ageing Res Rev. 2015 Mar;20:74-8. doi: 10.1016/j.arr.2014.10.003. Epub 2014 Oct 18. PMID 25461244
- [Background] Alhassan S, Kim S, Bersamin A, King AC, Gardner CD. Dietary adherence and weight loss success among overweight women: results from the A TO Z weight loss study. Int J Obes (Lond). 2008 Jun;32(6):985-91. doi: 10.1038/ijo.2008.8. Epub 2008 Feb 12. PMID 18268511
- [Background] Charan J, Biswas T. How to calculate sample size for different study designs in medical research? Indian J Psychol Med. 2013 Apr;35(2):121-6. doi: 10.4103/0253-7176.116232. PMID 24049221